CLINICAL TRIAL: NCT03064308
Title: The Assessment of the Feasibility of a Home Based Post-operative Exercise Training Programme Targeting Physical and Cognitive Function in Older Patients Undergoing Major Body Surgery
Brief Title: The Assessment of the Feasibility of a Home Based Exercise Programme in the Older Patient Following Major Surgery
Acronym: POETold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16014
Record Dates: First submitted 2016-02-25; First posted 2017-02-27 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2017-10

CONDITIONS: Impaired Cognition; Quality of Life; Surgery; Delirium; Colorectal Carcinoma; Bladder Carcinoma; Abdominal Hysterectomy (& Wertheim); Prostatic Neoplasms; Colon Carcinoma; Renal Carcinoma
Keywords: Frailty; Surgery; Physical function; Cognitive function; Quality of life; Exercise; Rehabilitation; Delirium; Morbidity; Mortality; Length of stay; Well-being; Elderly; Older surgical patient; Radical prostatectomy; Radical cystectomy; Radical cystoprostatectomy; Aortic Aneurysm Repair; Major Cavity Surgery; Abdominal Surgery; Recovery; Nephrectomy
MeSH Terms: conditions — Cognition Disorders; Delirium; Colorectal Neoplasms; Urinary Bladder Neoplasms; Prostatic Neoplasms; Colonic Neoplasms; Carcinoma, Renal Cell; Frailty; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will receive standard NHS care with no intervention.
- Exercise (Other): Participants will receive standard NHS care and complete the exercise programme, the intervention.
  Interventions: Other: Exercise Programme

INTERVENTIONS:
Other: Exercise Programme — Participants will complete the High-Intensity Functional Exercise (HIFE) programme. The programme improves lower-limb strength, balance and mobility and all the exercises can be performed by the individual at home and with minimal equipment.
  Arms: Exercise

SUMMARY:
The primary aim of this study is to establish if it is possible for patients who have undergone major body surgery to complete a home based exercise training program and complete the assessments required to measure physical and cognitive function. If the investigators can establish that it is feasible to complete the training and test's then further research can follow using these methods to determine whether it is possible to improve the physical function of older patients undergoing major abdominal surgery in the period following surgery by using a simple exercise regimen that can be carried out at home. By targeting physical function in this way the investigators hope to determine if it is a method for improving frailty and well being. In turn it may also have a positive impact on health service provision.

DETAILED DESCRIPTION:
Frailty is a geriatric syndrome describing a lack of physiological reserve. It is an independent risk factor for morbidity, mortality and increased length of hospital stay. Five criteria can be used to describe Frailty: weight loss, exhaustion, diminished hand-grip strength, slow walking speed, and low physical activity. Sarcopenia, the loss of skeletal muscle mass and strength, is a key component of all of these criteria and of Frailty itself.

By assessing Frailty, vulnerable patients can be recognised early so that additional measures can be implemented. Interventions to ameliorate the severity of an individual's Frailty are currently the focus of much attention as these can positively impact on the patients physical and cognitive function and well-being. In turn this has a positive impact on health service provision reducing hospital length of stay, morbidity and mortality.

The exercise programme used in this study incorporates the High-Intensity Functional Exercise (HIFE) programme for older individuals developed by Umea University Sweden with exercises incorporated from the Help the Aged Preventing Falls Programme. The exercises are designed such that they can be performed at home with no additional aids. The participants will be required to begin the programme on discharge from hospital and undertake exercises three times per week. They will receive instruction, help and support prior to discharge and throughout the 6 month exercise period. The participants will be required to complete an exercise diary to monitor their compliance with the programme and to determine the feasibility of a home based exercise programme as an intervention measure.

The outcome measures of physical function will be assessed by the Handgrip strength and Step Box testing plus questionnaires assessing daily activities, Sarcopenia will be assessed using the Handgrip test to measure muscle strength and quantification of muscle mass through muscle ultrasound (USS) imaging. Cognitive function will be assessed by the use of validated questionnaire and online cognitive tests. Frailty by the Reported Edmonton Frail Scale.

Experimental design and methods:

Potential participants will be identified from local multidisciplinary team (MDT) meetings. These are held weekly and all patients undergoing major cavity intra-abdominal surgery are discussed at the relevant MDT for their surgical speciality. Those patients who meet the eligibility criteria will be noted by the usual care team and they will make the initial approach to the patient regarding the study.

30 participants will be recruited to the study and allocated randomly to either the exercise intervention arm or the control arm of the study. Participants will be involved in the study for approximately 8 months depending upon when they are recruited to the study pre-operatively. The post-operative exercise programme runs for 6 months.

All aspects of the screening process are part of the standard NHS pre-operative assessment and include National Health Service (NHS) blood tests, ECG, clinical examination and medical questionnaire.

Participants will be asked to attend five testing sessions, one pre-operatively and four postoperatively. These sessions will wherever possible be timed with planned clinic appointments scheduled as part of the standard NHS care provided by their surgical speciality. The first session shall occur at the time of the pre-operative assessment and will require the participant to complete all of the assessments (detailed below). The second session occurs three days postoperatively whilst the participant is an inpatient, of the physical assessments only the handgrip strength test shall be completed. The remaining three sessions occur at 6 weeks, 3 months and 6 months post-operatively and all of the assessments shall be completed. At each session blood tests for monitoring of Haemoglobin levels and inflammatory markers shall be collected, some of which will be a part of the standard NHS care.

Assessment of physical function and Sarcopenia:

Handgrip test: Three readings (maximal isometric contraction of the hand using the Takei hand dynamometer) for each hand will be recorded with the average of the three readings calculated.

Step Box test: Participants will complete three sets of step box steps. The first set involves 10 steps at a slow pace, the second set, 20 steps at normal walking pace and the final set, 20 steps as fast as they can. The height of the step is dependent upon the height of the participant. The time to complete each set and the heart rate during stepping and in the recovery period is recorded.

The recovery period is 5 minutes or the time taken for the heart rate to return within 5 bpm of the resting heart rate.

Ultrasound of vastus lateralis: Ultrasound images will be taken of the vastus lateralis at a point 2/3 along the axis from the greater trochanter of the femur and the knee joint-line. At this point a sagittal image will be captured to delineate the anterior and posterior borders of the muscle. Muscle depth, bulk and muscle pennation angle will be calculated.

Assessment of Frailty:

Reported Edmonton Frail Scale: This is a validated frailty scoring system.

Assessment of Cognition:

The Montreal Cognitive Assessment (MoCA) questionnaire is a validated cognitive screening tool to screen for mild to moderate cognitive impairment.

Computerised Cognitive test battery: This involves two computerised tests, the Simon test and the Symbol Substitution test.

Questionnaires:

The following validated questionnaires will be used; The Duke Activity Status Index (DASI) assess activities of daily living, the EQ5D evaluates health status, the International Physical Activity - Short Form (IPAC-SF) questionnaire assess physical activity. Depression shall also be screened for by using the Geriatric Depression Scale (GDS).

Assessment of Feasibility:

The feasibility of the intervention will be determined through interviews, exercise diary's and feedback questionnaires.

Removal of participants from the study:

Patients will be withdrawn from the study if they wish to withdraw consent or loose the capacity to consent. Further if they develop post-operative complications of the cardio-vascular system, cerebrovascular system or complications of the operative wound site. Also if they discontinue with the exercise programme either temporarily or permanently.

Sample size calculation:

This is a feasibility study, there is no current data from which to estimate the sample size.

ELIGIBILITY:
* Inclusion Criteria:

  * Patients undergoing major body cavity surgery.
  * Male and Female patients.
  * Age greater than 70 years.
  * Patients undergoing neo-adjuvant chemotherapy will be included.
* Exclusion Criteria:

  * Participation in a formal exercise regime
  * A BMI > 35 kg·m2
  * Active cardiovascular disease: uncontrolled hypertension (BP > 180/100), angina, heart failure (class III/IV), arrhythmia, right to left cardiac shunt, recent cardiac event
  * Taking beta-adrenergic blocking agents.
  * Cerebrovascular disease: untreated aneurysm (large vessel or intracranial).
  * Respiratory disease including: pulmonary hypertension.
  * Metabolic disease: hyper and hypo parathyroidism, untreated hyper and hypothyroidism, Cushing's disease.
  * Musculoskeletal or neurological disorders
  * Family history of early (<55y) death from cardiovascular disease
  * Severe rheumatoid arthritis limiting ability to perform any part of the assessment process.
  * Unable to complete the consent process.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Feasibility of a home based exercise programme following surgery in the older patient. | 3 and 6 months
  To determine the feasibility of a post-operative home based exercise program at 3 and 6 months, for older patients over 70 years of age, who have undergone major body cavity surgery. To assess if this approach is an acceptable and practically viable health intervention in this demographic group. The feasibility will be assessed through the use of interviews with the participants, review of the participants exercise diary and written participant feedback.

SECONDARY OUTCOMES:
Step Box Test | 3 and 6 months
  The difference in estimated maximal oxygen consumption (VO2 max) pre-operatively (baseline) and post-operatively at 3 months and 6 months following a post-operative exercise training programme.
Muscle Architecture Ultrasound | 3 and 6 months
  The assessment of lean muscle architecture using ultrasound techniques. Muscle fibre length and pennation angle will be measured and compared pre-operatively (baseline) and post-operatively at 3 months and 6 months following a post-operative exercise training programme.
Cognitive testing | 3 months
  Cognition shall be compared pre-operatively (baseline) and at 3 months and 6 month post-operatively through completion of the Montreal Cognitive Assessment questionnaire and the utilisation of computerised cognitive testing programmes to assess the effect of a post-operative exercise training programme. The results of the cognitive tests shall be pooled to provide an overall cognitive outcome measure.
Frailty | 3 and 6 months
  Frailty scores using the Reported Edmonton Frail Scale shall be compared pre-operatively (baseline) and post-operatively at 3 months and 6 months following a post-operative exercise training programme
Subjective Outcome measure: Physical Activity. | 3 and 6 months
  The Duke Activity Status Index (DASI) measures physical activity. This in conjunction with the other subjective outcomes will enable a overview of quality of life to be made. The questionnaire will be completed at 3 and 6 months.
Subjective Outcome measure: VO2max measure | 3 and 6 months
  The Duke Activity Status Index (DASI) will measure VO2max. This in conjunction with the other subjective outcomes will enable a overview of quality of life to be made. The questionnaire will be completed at 3 and 6 months.
Subjective Outcome measure: Physical Activity | 3 and 6 months
  The International Physical Activity Questionnaire (IPAC-SF) will measure the nature of the physical activity taken place and time dedicated to this. This questionnaire is designed and validated for the older population. This questionnaire in conjunction with the other subjective outcomes will enable a overview of quality of life to be made. The questionnaire will be completed at 3 and 6 months.
Subjective Outcome measure: Quality of Life | 3 and 6 months
  The EQ-5D-3L is a validated questionnaire measuring quality of life. This questionnaire in conjunction with the other subjective outcomes will enable a overview of quality of life to be made. The questionnaire will be completed at 3 and 6 months.
Hand Strength Test | 3 and 6 months
  The difference in hand strength measurements pre-operatively (baseline) and post-operatively at 3 and 6 months following a post-operative exercise training programme.

OTHER OUTCOMES:
Intervention Compliance Questionnaire | 3 and 6 months
  Patient compliance and adherence to training programs at 3 and 6 months post-operatively assessed subjectively by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: John Williams, MBChB PhD, Study Chair — Clinical Associate Professor and Consultant Anaesthetist; Bethan Phillips, BSc PhD, Study Director — Assistant Professor; Jon Lund, MD, Study Director — Clinical Associate Professor and Consultant Colorectal Surgeon; Laura Carrick, BSc MBChB, Principal Investigator — Clinical Research Fellow, Specialist Registrar in Anaesthetics
Locations (1):
- Division of Graduate Entry Medicine and Health, School of Medicine, University of Nottingham. Royal Derby Hospital,, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No